CLINICAL TRIAL: NCT00094484
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of Cinacalcet HCl in Chronic Kidney Disease Subjects With Secondary Hyperparathyroidism Not Receiving Dialysis
Brief Title: Cinacalcet HCl in Chronic Kidney Disease Subjects With Secondary Hyperparathyroidism Not Receiving Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 20000178
Record Dates: First submitted 2004-10-19; First posted 2004-10-20 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Kidney Disease; Chronic Kidney Disease
Keywords: Sensipar®; Mimpara®; Cinacalcet; Calcimimetic; Chronic Kidney Disease
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic | interventions — Cinacalcet

INTERVENTIONS:
Drug: Cinacalcet HCl

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of cinacalcet compared with placebo in patients with stage 3 and 4 Chronic Kidney Disease (CKD).

ELIGIBILITY:
Inclusion Criteria: Chronic Kidney Disease patients not receiving dialysis with: - An iPTH greater than 100 pg/mL [10.6 pmol/L] for subjects with stage 3 CKD or greater than or equal to 160 pg/mL [17.0 pmol/L] for subjects with stage 4 CKD; - A serum calcium greater than 9.0 mg/dL [2.25 mmol/L]; - An estimated GFR less than or equal to 59 mL/min and greater than or equal to 15 mL/min. Exclusion Criteria: - Have an unstable medical condition, defined as having been hospitalized within 30 days before day 1, or otherwise unstable in the judgment of the investigator. - Experienced a myocardial infarction (MI) within 3 months before day 1. - Likely to initiate dialysis (in the opinion of the investigator) or are scheduled to undergo renal transplantation within 28 weeks after day 1. - Received active vitamin D therapy (i.e., 1-hydroxylated metabolites of vitamin D) for less than 30 days before day 1 or required a change in active vitamin D brand or dose level within 30 days before day 1 (for patients prescribed active vitamin D).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2004-10

PRIMARY OUTCOMES:
Proportion of subjects with a mean reduction of greater than or equal to 30% in iPTH at 32 weeks

SECONDARY OUTCOMES:
Changes in iPTH at 32 weeks.
Safety and tolerability of cinacalcet at 32 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Chonchol M, Locatelli F, Abboud HE, Charytan C, de Francisco AL, Jolly S, Kaplan M, Roger SD, Sarkar S, Albizem MB, Mix TC, Kubo Y, Block GA. A randomized, double-blind, placebo-controlled study to assess the efficacy and safety of cinacalcet HCl in participants with CKD not receiving dialysis. Am J Kidney Dis. 2009 Feb;53(2):197-207. doi: 10.1053/j.ajkd.2008.09.021. Epub 2008 Dec 24. PMID 19110359
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_38_AMG_073_20000178.pdf
- See also: FDA-approved Drug Labeling — http://www.sensipar.com/